CLINICAL TRIAL: NCT07123480
Title: The Impact of Informed Consent Type on Participation in an Implementation Science Pilot Study to Improve Cardiac Rehabilitation Participation
Brief Title: The Role of 4 Different Consent Approaches on a Pilot Study to Increase Cardiac Rehabilitation Attendance
Acronym: MOST-CR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baystate Medical Center (Other)
Responsible Party: Principal Investigator, Quinn Pack, MD, MSc, Medical Director of Cardiac Rehabilitation and Wellness, Baystate Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2311694
Record Dates: First submitted 2025-08-04; First posted 2025-08-14 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Ethics; Cardiac Rehabilitation; Coronary Heart Disease (CHD); Heart Failure; Percutaneous Coronary Intervention (PCI); Aortic Valve Replacement; Myocardial Infarction (MI)
Keywords: Cardiac Rehabilitation; Informed Consent Approach; Phase 2; implementation science
MeSH Terms: conditions — Coronary Disease; Heart Failure; Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: An open-label prospective double randomized control study at Baystate Medical Center, a 760-bed academic teaching hospital. Patients are first randomized to one of the four consent approaches. If the patients agree to participate or are in the non-consent group, the patients will be re-randomized 1:1 to either Usual Care or the More Support and Tools Program (MOST).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Long Consent (Other): Standard Consent approach (typically 10-12 pages)
  Interventions: Behavioral: Usual Care Group; Behavioral: More Support and Tools
- Short Consent (Other): Three page key Information consent
  Interventions: Behavioral: Usual Care Group; Behavioral: More Support and Tools
- Opt-Out (Other): 1 page opt-out consent approach
  Interventions: Behavioral: Usual Care Group; Behavioral: More Support and Tools
- Non-Consenting (Other): No consent
  Interventions: Behavioral: Usual Care Group; Behavioral: More Support and Tools

INTERVENTIONS:
Behavioral: Usual Care Group — Standard of care to encourage cardiac rehabilitation attendance.
Behavioral: More Support and Tools — More Support and Tools includes the following: monetary incentive, text messages, case management, and physical activity coaching. The investigators will start providing support and tools while patients are still in the hospital and continue this support weekly after discharge. Intervention participants will receive a monetary incentive both in the hospital and upon attending cardiac rehabilitation. The support (case management) and tools (physical activity coaching and text messages) will continue for up to 3 months or until the individual attends cardiac rehabilitation, whichever occurs first. Participants can decline any or all support or tools.

SUMMARY:
Cardiac Rehabilitation is a lifestyle and exercise program for patients with heart disease. Cardiac Rehabilitation is strongly recommended in guidelines, but only 30% of eligible patients attend.

New strategies are needed to help more patients attend cardiac rehabilitation. In this study, the investigators will see if using an $50 incentive, case management, text messages, and physical activity coaching combined into a single intervention will help more patients attend cardiac rehabilitation.

In preparation for a larger trial, patients will also be randomly assigned to four different ways of seeking their permission to be in a research study. The investigators will see if these approaches affect how many people participate in the research project.

The two main goals of this study is to understand:

1. If the consent approach type impacts participation rates in the research study
2. If the multi-component intervention (case management, financial incentives, text messages, and physical activity coaching) improves cardiac rehabilitation participation within 3 months.

DETAILED DESCRIPTION:
Cardiac Rehabilitation (CR) is a guideline-recommended therapy that helps patients improve their health and longevity. It is underused, especially among older, sicker, and minority populations. Guidelines make strong recommendations for use among all patients, and there are ongoing national initiatives to improve utilization. At Baystate, cardiac rehabilitation attendance rates are improving, but investigators are still seeking additional strategies to further encourage participation. If the investigators succeed, patients will live longer, healthier lives, thus embodying beneficence.

However, the typical 10-12 page consent form is a major barrier to successful study completion with participation rates in typical clinical trials of 20% of eligible patients. More importantly, it introduces an important selection bias in the population by finding patients who are more responsive to interventions. It also shifts the population towards patients away from underrepresented minorities and yields results that are less applicable to real-world settings with clinical populations. In short, this selection bias is inconsistent with the ethical principle of justice, which states that the same population that is expected to benefit from the research should also be the population that bears the burden of the research. Thus, alternate forms of informed consent are needed to assure a representative population and scientific results that can be confidently generalized.

First, to address issues of consent, the investigators will determine the impact of four different ethical approaches to consent (full consent with signature, 3-page summary consent with signature, 1-page opt-out waiver - no signature, or Non-Consenting (NC) cohort - where patients can refuse any intervention) on study enrollment rate and population representativeness.

Second, the investigators will assess the feasibility and utilization of a multi-dimensional intervention to increase CR enrollment. These will include combining a financial incentive, case management, text messaging program, and physical activity coaching, all with the goal of increasing CR enrollment. The investigators will assess the acceptance rate of intervention components and the overall feasibility of the proposed intervention in preparation for larger clinical trials.

Patients will be randomized to 1 of 4 consent approaches shown below. All consent documents and corresponding waivers were submitted to a full board IRB and approved.

* Full consent form. This is the typical 10 to 12-page consent form at Baystate Medical Center. This has the 3-4-page summary and the 6-8 pages of technical details. It has unalterable language provided by the Baystate Institutional Review Board (IRB) and Baystate Legal with an 11th-grade Keiser-Fleischer reading grade level. All elements of consent are included. A full HIPPA waiver is included. Signature is required.
* Brief consent form. This 3-4-page consent form summarizes the study in a shorter form. All essential information is retained, and there is considerably less required legal language. Signature is required. The investigators provided a justification for alteration of consent to our IRB.
* 1 page opt-out Waiver. This 1-page description includes a brief description of the study, its purposes, and goals. It gives the patient a chance to opt-out, but does not require a signature. Patients' consent is implied unless they indicate otherwise. The investigators provided a justification for alteration of consent to their IRB.
* Non-Consenting (NC) Cohort. Patients are told they are participating in a Cardiac Rehabilitation Project, but are given the option to decline any intervention they are not interested in. The investigators will not provide written or explicit verbal consent prior to participating. The investigators provided a Justification for alteration of consent to their IRB.

Patients who agree to participate by signing a consent form, by not opting out, or by being randomized to the non-consent group will be re-randomized to either the Usual Care or MOST group. Additional details of these interventions are found below.

If patients consent, do not opt-out, or are randomized to the non-consenting cohort, they will be re-randomized 1:1 to either usual care or a multifactorial CR intervention. This intervention will include four components: financial incentives, text messaging, case management, and physical activity coaching, combined as a single intervention.

The primary outcome will be the proportion of patients (%) participating in the clinical trial. The secondary outcome will be enrollment in CR within 3 months of hospital discharge.

All interventions are minimal risk. They are typically found in routine clinical medicine and have been used without difficulty in other settings. In any group, patients can refuse any or all components of the intervention, thus respecting patient autonomy. If patients respond and attend CR, they will gain health benefits, which is consistent with the ethical principle of beneficence.

ELIGIBILITY:
Inclusion Criteria:

* Only Baystate Medical Center (Springfield, Massachusetts ) adult patients over age 18 who are admitted to Baystate Medical Center Hospital with a non-surgical qualifying diagnosis for outpatient CR will be included. Common diagnoses include all patients with myocardial infarction, stable angina, percutaneous coronary intervention, transcutaneous aortic/mitral valve replacement, and heart failure.

Exclusion Criteria:

- Patients with coronary artery bypass graft surgery, heart valve surgery, or other open-heart surgical procedures will be excluded, as these patients are much more likely attend CR, typically around 70%. In addition, patients who are referred to CR programs outside the region, where enrollment cannot be tracked, will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Informed Consent Approach Participation | Baseline
  The proportion of patients (%) participating in the clinical trial.

SECONDARY OUTCOMES:
Cardiac Rehabilitation Attendance | Up to to 3 months after hospital discharge, or cardiac rehabilitation attendance, whichever comes first.
  The proportion (%) of patients who attend 1 or more sessions of cardiac rehabilitation
Age Representativeness of Consenting Groups | Baseline
  Each consent group will be analyzed based on the demographics of patients participating. The age characteristics of each consent group will be measured in years.
Sex Representativeness of Consenting Groups | Baseline
  Each consent group will be analyzed based on the demographics of patients participating. The sex characteristics of each consent group will be measured as male, female, or other.
Race Representativeness of Consenting Groups | Baseline
  Each consent group will be analyzed based on the demographics of patients participating. The race characteristics of each consent group will be measured using the five NIH racial categories (American Indian or Alaska Native, Asian, Black or African American, Native Hawaiian or Other Pacific Islander, and White).
Ethnicity Representativeness of Consenting Groups | Baseline
  Each consent group will be analyzed based on the demographics of patients participating. The ethnicity characteristic of each consent group will be measured using the NIH defined categories (Hispanic or Latino, and Not Hispanic or Latino).
Cardiac Rehabilitation Qualifying Diagnosis Representativeness of Consenting Groups | Baseline
  Each consent group will be analyzed based on the demographics of patients participating. The cardiac rehabilitation qualifying diagnosis characteristic of each consent will be measured.
The Porportion of Intervention Accepted | Up to to 3 months after hospital discharge, or cardiac rehabilitation attendance, whichever comes first
  The proportion of patients (%) who accept each intervention (financial incentives, case management, physical activity coaching, and text messaging) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Quinn R Pack, MD, MSc, Principal Investigator — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual data may be shared, but given that patients are randomized to 4 different informed consent approaches, one of which is a non-consent group, it is unclear if the Institutional Review Board (IRB) would allow data sharing. At this time, data sharing seems unlikely.